CLINICAL TRIAL: NCT03886103
Title: Pharmacokinetics and Metabolism of [14C]-Labelled PXL770 Following a Single Oral Administration in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Metabolism of (14C)-Labelled PXL770
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXL770-005
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteer (Experimental): Single of 14C-PXL770
  Interventions: Drug: 14C labeled PXL770

INTERVENTIONS:
Drug: 14C labeled PXL770 — Single administration

SUMMARY:
This is a single-dose, single center, single-period, open-label, non-randomized, mass balance recovery study in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males
* Age 30 to 65 years
* BMI 18.5 to 32.0 kg/m2 and body weight of 55 to 95 kg.
* Must be willing and able to communicate and participate in the whole study
* Must have regular bowel movements (ie, average stool production of ≥1 and ≤3 stools per day)
* Must provide written informed consent
* Regular alcohol consumption of 4-14 units of alcohol per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
* Must agree to adhere to the contraception

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the previous 3 months or 90 days prior to Day 1
* any drug or alcohol abuse
* Current smokers and those who have smoked within the last 12 months.
* Radiation exposure, including that from the present study, excluding background adiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years.
* No occupationally exposedworker, as defined in the Ionizing Radiation Regulations 2017, shall participate in the study
* Clinically significant abnormal biochemistry, hematology, coagulation or urinalysis as judged by the investigator
* Positive test for HIV, HBV, HBC
* eGFR <80 mL/min
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or GI disease, neurological or psychiatric disorder, as judged by the investigator
* Known sensitivity to any of the constituents or excipients of the study drug or history of relevant drug and/or food allergy (anaphylactic, anaphylactoid reactions)
* History of drug-induced Torsade de Pointe or presence of a familial long QT syndrome
* Mental handicap

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery | From day 1 to day 7
  Mass balance recovery of total radioactivity in all excreta: cumulative recovery (CumAe) and cumulative recovery expressed as a percentage of the dose (Cum%Ae)

SECONDARY OUTCOMES:
PK profile of total radioactivity | From day 1 to day 7
  Cmax
PK profile of PXL770 | From day 1 to day 7
  Cmax
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From day 1 to day 7
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient, Nottingham, United Kingdom